CLINICAL TRIAL: NCT02984215
Title: Array-CGH in Plasma Cell Post-transplantation Lymphoproliferative Disorders
Brief Title: aCGH Impacts Survival in Plasma Cell PTLD
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL16_0720
Record Dates: First submitted 2016-10-31; First posted 2016-12-06 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-10

CONDITIONS: Post-transplantation Lymphoproliferative Disorders

STUDY DESIGN:
Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — the investigators report array-based comparative genomic hybridization (aCGH) of 10 cases of PCM and PLL-PTLD. aCGH performed on 10 plasma cell PTLD.

SUMMARY:
Plasma-cell post-transplantation lymphoproliferative disorders (PC-PTLD) are rare monomorphic PTLD divided into plasma cell myeloma (PCM) and plasmacytoma-like lesion (PLL) PTLD. To date, there is no exhaustive published cytogenetic data on PC-PTLD. The investigators report array-based comparative genomic hybridization (aCGH) of 10 cases of PCM and PLL-PTLD.

ELIGIBILITY:
Inclusion Criteria:

* WHO classification 2008 as monomorphic PCM (plasma cell myeloma) or PLL (plasmacytoma like lesion) / PTLD (post transplantation lymphoproliferative disorders).

Exclusion Criteria:

* Other than PCM or PLL PTLD at diagnosis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: We conducted a retrospective analysis between 1990 and 2012 of all consecutive cases of PCM and PLL-PTLD collected in the Centre Hospitalier Lyon Sud (CHLS, 6 cases) and in Necker - Enfants Malades Hospital in Paris (4 cases). There were 4 females and 6 males. Among the 8 adults, 6 had received a kidney transplant, 1 a heart transplant and one a lung transplant. Among the 2 children, one had received a heart transplant and one an allogeneic stem cell transplantation with a matched unrelated donor. Immunosuppressive regimens were heterogeneous.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 1990-01; Primary Completion 2012-01 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Genome wide array-based comparative genomic hybridization (aCGH) | At diagnosis of PTLD, Day 0.

SECONDARY OUTCOMES:
Overall survival according to aCGH complexity | Overall survival (OS) was calculated from date of diagnosis to date of death from any cause, up to 130 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre hospitalier Lyon sud, Pierre-Bénite, Auvergne-Rhône-Alpes, France